CLINICAL TRIAL: NCT01241526
Title: An International Phase IV Randomised Trial for Medical and Medico-economic Evaluations of Home-based Disease Management Program in Patients With Gold III/IV Chronic Obstructive Pulmonary Disease.
Brief Title: The COPD Patient Management European Trial (COMET)
Acronym: COMET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Collaborators: ITEC Services (Other); Lincoln Medical and Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ALMED-07-C4-008
Record Dates: First submitted 2010-11-09; First posted 2010-11-16 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; COMET; Disease management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Disease Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Disease management program (Experimental)
  Interventions: Other: Disease Management
- Usual site management (Active Comparator)
  Interventions: Other: Usual site management

INTERVENTIONS:
Other: Disease Management — * Individual, group and phone education sessions
  * Telephone supporter follow-up
  * LTOT monitoring
  Other Names: Living Well With COPD Disease Management Program
  Arms: Disease management program
Other: Usual site management — * Usual education as per site protocol
  * Usual follow-up as per site protocol
  * LTOT monitoring
  Arms: Usual site management

SUMMARY:
The goal of the study is to evaluate a Home-Based Disease Management program specifically developed for patients with Gold III/IV COPD.

By improving disease knowledge, awareness of significant clinical deterioration and self-management skills for patients, this Home-Based COPD Management Program is expected to reduce the severity of exacerbations, the need for emergency hospitalisations, thus demonstrating the efficacy and the cost effectiveness of this intervention.

DETAILED DESCRIPTION:
Primary objective: To evaluate a strategy of Chronic Obstructive Pulmonary Disease (COPD) management to reduce the number of hospital days in patients with severe Gold III/IV COPD: a Home-Based COPD Management Program versus usual patient education and follow-up.

Secondary objectives:

* To assess the clinical outcome and the health-related quality of life,
* To assess safety,
* To evaluate medico-economic impact.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Gold III/IV COPD
* Current or ex-smoker with a smoking history ≥ 10 pack-years
* At least one COPD exacerbation leading to hospitalization in the year before selection.

Exclusion Criteria:

* LTOT for another reason than COPD
* Severe concomitant disorder associated with a limited probability of survival (< 6 months)
* Tracheostomy
* Long term oral corticosteroids therapy

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2010-09; Primary Completion 2015-02 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of unscheduled hospital days | up to 12 months

SECONDARY OUTCOMES:
Number of hospital days due to severe COPD exacerbation | up to 12 months
Safety parameters | up to 12 months
  Adverse Events (AEs)
Medico-economic data | up to 12 months
  Cost estimation, Cost-effectiveness, Cost-utility.
Health related quality of life | up to 12 months
Use of health care services | up to 12 months
Compliance to oxygen therapy | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Romain KESSLER, MD, Study Chair — Hopital Civil de Strasbourg - France
Locations (34):
- France (13):
  - Centre Hospitalier d Antibes Juans-les-pins, Antibes
  - Hôpitaux Civils de Colmar - Hôpital Pasteur, Colmar
  - CHU de Grenoble, Grenoble
  - Centre Hospitalier du Mans, Le Mans
  - Hôpital de la Croix Rousse, Lyon
  - Assistance Publique Hôpitaux de Marseille - Hôpital Nord, Marseille
  - Hôpital MERCY, Metz
  - Hôpital Saint Louis, Paris
  - Groupe Hospitalier Pitié-Salpétrière, Paris
  - Groupe Hospitalier Saint Joseph, Paris
  - Hôpital Civil de Strasbourg, Strasbourg
  - Hôpital Beauregard - CHR METZ, Thionville
  - Hôpital Sainte Musse, Toulon
- Germany (8):
  - Marien Krankenhaus, Kassel, Hesse
  - Universitatklinikum, Aachen
  - Helios Hagen-Ambrock, Hagen
  - Thoraxklinik Heidelberg gGmbh, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Fachkrankenhaus Kloster Grafschaft, Schmallenberg
  - Klinik für Pneumologie und Allergologie, Solingen
  - Universitätsklinikum Ulm, - Klinik Innere Medizin II, Ulm
- Italy (6):
  - Azienda ULSS 22 - Ospedale di Bussolengo, Bussolengo
  - ASL Viterbo, Civita Castellana
  - Ospedale di Macerata, Macerata
  - Azienda Ospedaliera, "Ospedale San Carlo Borromeo", Milan
  - "Azienda Ospedaliera Niguarda, Milan
  - Azienda ospedialiera Di DESIO Vimercate, Seregno
- Spain (7):
  - Hospital La Princessa, Madrid, Madrid
  - Hospital Gregorio Maranon, Madrid, Madrid
  - Hospital Ramon Y Cajal, Madrid, Madrid
  - Hospital Universitario de Burgos, Burgos
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario de Asturia, Oviedo
  - Hospital Arnau de Vilanova, Valencia

REFERENCES:
- [Derived] Poot CC, Meijer E, Kruis AL, Smidt N, Chavannes NH, Honkoop PJ. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Sep 8;9(9):CD009437. doi: 10.1002/14651858.CD009437.pub3. PMID 34495549
- [Derived] Kessler R, Casan-Clara P, Koehler D, Tognella S, Viejo JL, Dal Negro RW, Diaz-Lobato S, Reissig K, Rodriguez Gonzalez-Moro JM, Devouassoux G, Chavaillon JM, Botrus P, Arnal JM, Ancochea J, Bergeron-Lafaurie A, De Abajo C, Randerath WJ, Bastian A, Cornelissen CG, Nilius G, Texereau JB, Bourbeau J. COMET: a multicomponent home-based disease-management programme versus routine care in severe COPD. Eur Respir J. 2018 Jan 11;51(1):1701612. doi: 10.1183/13993003.01612-2017. Print 2018 Jan. PMID 29326333